CLINICAL TRIAL: NCT06640010
Title: Using Induced-Pluripotent Stem Cells to Model Cancer Therapy-Related Adverse Events
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC240101; NCI-2024-08355 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-002830 (Other: Mayo Clinic Institutional Review Board); MC240101 (Other: Mayo Clinic)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to find out if patient blood samples can be used to perform individualized modeling of cancer therapy-related side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Generate induced pluripotent stem cells (iPSC's) from patients receiving cancer treatment.

II. Differentiate patient iPSC's into cardiomyocytes and/or neurons or other cell types that may be relevant to modeling cancer therapy-related adverse effects, such as cardiotoxicity and neurotoxicity.

III. Use patient specific iPSC-derived cells to:

IIIa. Model cancer therapy-related toxicities; IIIb. Better understand the mechanisms of toxicities; IIIc. Determine if patient specific genetic variants are causative of toxicities; IIId. Screen novel protective therapies for cancer therapy-related toxicities.

OUTLINE: This is an observational study.

Patients undergo blood sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient >= 18 years of age
* Previously treated, planned or currently receiving any potentially toxic cancer therapy including but not limited to chemotherapy, targeted and immunotherapies

Exclusion Criteria:

* Inability on the part of the patient to understand the informed consent or be compliant with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients who have already started or are planning to start cancer treatment
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
In vitro measurement of cellular viability in response to chemotherapy | Blood drawn at enrollment to obtain sample
  Will be compared between cells derived from patients who experienced treatment-induced toxicity to cells derived from patients who received the same cancer therapy without toxicity. Statistical analyses of different endpoints will use Fisher's exact test, one-way ANOVA test followed by all-pairwise-multiple-comparison procedures, or an unpaired, two-tailed Student's t-test with significant differences defined by P < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Norton, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials